CLINICAL TRIAL: NCT05397912
Title: Uterine Elastography: a Potential Predictor of Embryo Transfer Success
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2022-02
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women undergoing euploid, single frozen embryo transfer: Women age 18yo-45yo undergoing euploid, single, frozen embryo transfer with sonographically normal appearing uterus without uterine factor infertility
  Interventions: Diagnostic Test: Uterine Elastography

INTERVENTIONS:
Diagnostic Test: Uterine Elastography — Shear wave elastography data will be obtained at the transvaginal ultrasound visit the day prior to frozen embryo transfer

SUMMARY:
To determine if the mean elasticity value (measured in kilopascals, kPa) of a patient's endometrium, myometrium and cervix in a sonographically normal appearing uterus predict frozen embryo transfer (FET) success and long term reproductive outcomes when measured the day prior to FET.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, 18yo-45yo, presenting for ultrasound the day prior to embryo transfer
2. Patients planning to undergo single embryo transfer (SET) of a euploid embryo by Preimplantation genetic testing for aneuploidy (PGT-A)
3. Uterine evaluation prior to transfer (saline sonogram or hysteroscopy) within 1 year
4. Egg recipients

Exclusion Criteria:

1. Gestational carriers
2. BMI > 35
3. Diagnosis of a uterine anomaly
4. History of uterine surgery, excluding polypectomy, c-section, D&C
5. Communicating hydrosalpinx
6. Transfer of an embryo of unknown ploidy status or embryos of undetermined safety
7. Surgically retrieved sperm
8. Embryos that were cryopreserved on day 7 of development
9. Poor quality embryos defined by modified Gardner grading criteria used in the embryology lab
10. Sonographically abnormal appearing uteri, including distortions from leiomyomas and thin endometrium

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients presenting to one of our offices for an ultrasound the day prior to embryo transfer will be reviewed for inclusion. Patients will be undergoing euploid, single, frozen embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Sustained Implantation Rate | 6 weeks after embryo transfer
  number of fetal heart beats at time of discharge ultrasound

SECONDARY OUTCOMES:
Chemical Pregnancy | 8-10 days after embryo transfer
  Positive serum bHCG level
Clinical Pregnancy | 2-4 weeks after embryo transfer
  presence of gestational sac on ultrasound
Clinical Pregnancy Loss | 2-40 weeks after embryo transfer
  loss of gestational sac, yolk sac, fetal pole, fetal heart beat on ultrasound after being present

CONTACTS AND LOCATIONS:
Overall Officials: Marie Werner, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Margolis C, Garrido N, Roberts L, Reig A, Gill P, Willson S, Genovese H, Barrett F, Zuckerman C, Whitehead C, Bergh P, Seli E, Werner M. Mapping the way to successful euploid frozen embryo transfer: a prospective pilot study of uterine elastography. Hum Reprod. 2025 May 1;40(5):895-903. doi: 10.1093/humrep/deaf029. PMID 39999405